CLINICAL TRIAL: NCT01109121
Title: A Randomized, Double-Blind, Parallel Group Study to Evaluate the Safety and Efficacy of Tranilast in Combination With Allopurinol in Patients With Moderate to Severe Gout (TAnGO)
Brief Title: Tranilast Plus Allopurinol in Patients With Moderate to Severe Gout (TAnGO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nuon Therapeutics, Inc. (Industry)
Responsible Party: Nuon Therapeutics Clinical Trials Contact, Nuon Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3007GT
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Moderate to Severe Gout; Hyperuricemia
Keywords: Moderate to severe gout; Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Allopurinol (Active Comparator): Allopurinol
  Interventions: Drug: Allopurinol
- Combination 400 (Experimental): Tranilast and Allopurinol
  Interventions: Drug: Combination 400
- Combination 600 (Experimental): Tranilast and Allopurinol
  Interventions: Drug: Combination 600

INTERVENTIONS:
Drug: Combination 400 — Tranilast 300 mg QD; Allopurinol 400 mg QD
  Arms: Combination 400
Drug: Allopurinol — Allopurinol 400 mg, QD
  Arms: Allopurinol
Drug: Combination 600 — Tranilast, 300 mg QD; Allopurinol 600 mg QD
  Arms: Combination 600

SUMMARY:
This Phase 2 study will be a multicenter, double-blind, randomized, active-comparator study to evaluate the safety and efficacy of tranilast in combination with allopurinol in patients with hyperuricemia and moderate to severe gout.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 80
* Severe gout, demonstrated by 3 or more gout flares in the previous 12 months, or the presence of at least one gout tophus or gouty arthritis
* Hyperuricemia with a sUA ≥8.0 mg/dL

Exclusion Criteria:

* Pregnant or nursing
* Known hypersensitivity to any of the components of tranilast or allopurinol
* Known history of xanthinuria or kidney stones
* Use of an investigational drug within 30 days
* Presence of, or history of, cancer with the exception of completely excised, non-metastatic squamous cell and basal cell carcinomas of the skin
* Subject is planning or likely to require a surgical procedure during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in serum uric acid (sUA) levels | 4 weeks

SECONDARY OUTCOMES:
Proportion of subjects whose sUA levels fall below 6.0 mg/dL following 4 weeks of dosing | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Director, Nuon Clinical Trials Group, Study Director — Nuon Therapeutics, Inc.
Locations (24):
- United States (24):
  - Nuon Investigative Site, La Jolla, California
  - Nuon Investigative Site, Santa Maria, California
  - Nuon Investigative Site, Washington D.C., District of Columbia
  - Nuon Investigative Site, New Port Richey, Florida
  - Nuon Investigative Site, Honolulu, Hawaii
  - Nuon Investigative Site, Boise, Idaho
  - Nuon Investigative Site, Bloomington, Indiana
  - Nuon Investigative Site, Owensboro, Kentucky
  - Nuon Investigative Site, Baltimore, Maryland
  - Nuon Investigative Site, Wheaton, Maryland
  - Nuon Investigative Site, Billings, Montana
  - Nuon Investigative Site, Omaha, Nebraska
  - Nuon Investigative Site, Reno, Nevada
  - Nuon Investigative Site, Teaneck, New Jersey
  - Nuon Investigative Site, Durham, North Carolina
  - Nuon Investigative Site, Cincinnati, Ohio
  - Nuon Investigative Site, Oklahoma City, Oklahoma
  - Nuon Investigative Site, Lake Oswego, Oregon
  - Nuon Investigative Site, Duncansville, Pennsylvania
  - Nuon Investigative Site, West Reading, Pennsylvania
  - Nuon Investigative Site, Charleston, South Carolina
  - Nuon Investigative Site, Greenville, South Carolina
  - Nuon Investigative Site, Waco, Texas
  - Nuon Investigative Site, Spokane, Washington